CLINICAL TRIAL: NCT00955799
Title: A Randomized, Double-Blind, Placebo-Controlled, Clinical Evaluation of the Efficacy, Safety and Tolerability of Neramexane in Patients With Subjective Tinnitus
Brief Title: Efficacy, Safety, Tolerability of Neramexane in Patients With Subjective Tinnitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRZ 92579/TI/3003; 2009-011246-25 (EudraCT Number)
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Subjective Tinnitus
Keywords: Subjective, Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neramexane mesylate (Experimental): Double-blind treatment period of 29 weeks up to 75 mg Neramexane mesylate per day
  Interventions: Drug: Neramexane mesylate
- Placebo (Placebo Comparator): Placebo: identical placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neramexane mesylate — Double-blind treatment period of 29 weeks up to 75 mg Neramexane mesylate per day
  Arms: Neramexane mesylate
Drug: Placebo — Double-blind treatment period of 29 weeks placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of neramexane mesylate in the treatment of subjective tinnitus in comparison to placebo.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients aged between 18 and 75 years with a clinical diagnosis of first onset, persistent (i.e., tinnitus should never be absent for > 24 hours in a row), subjective, uni- or bilateral subacute tinnitus

Main Exclusion Criteria:

* Clinical diagnosis of intermittent or pulsatile tinnitus
* Patients who have tinnitus as a concomitant symptom of an otological/neurological disease (such as otitis media, Menière's disease, otosclerosis, etc)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Absolute Change in TBF-12 (Tinnitus Handicap Inventory-12) Total Score from Baseline. | Baseline to week 17 and 29
  The TBF-12 is an adapted German version of the original English THI (Tinnitus Handicap Inventory). It is a self-report questionnaire assessing 12 items from 2 dimensions: emotional-cognitive factors and functional-communicational factors. Each item is rated with 0-2 (2= "often"; 1= "sometimes"; 0= "never"). The maximum score is 24 indicating most severe tinnitus impairment.
  Hierarchical test procedure: Step 1: week 29 in subjects reporting acute hearing loss; step 2: week 17, ditto; step 3: week 29 in total population; step 4: week 17, ditto.
Absolute Change in TSSw (Tinnitus Severity Scale - One Week Version) Total Score from Baseline. | Baseline to week 17 and 29
  The TSSw is a measure of tinnitus severity. It will be self-evaluated by the patient at various time points on an 11-point Likert-like scale asking for the past week. The scores range from 0 (indicating no tinnitus) to the maximum score of 10 (characterizing the most severe tinnitus considered).
  Hierarchical test procedure: Step 1: week 29 in subjects reporting acute hearing loss; step 2: week 17, ditto; step 3: week 29 in total population; step 4: week 17, ditto.

SECONDARY OUTCOMES:
TBF-12 Total Score: Change from Baseline | Baseline to week 5, 17, 23, and 29
  See outcome measure #1.
TBF-12 Factorial Scores: Change from Baseline | Baseline to week 5, 17, 23, and 29
  See outcome measure #1.
TBF-12: Individual Responder Rate | Week 5, 17, 23, and 29
  See outcome measure #1. A subject is considered responder if TBF-12 decreases at least 4 score points between baseline and respective visit.
Tinnitus Rating Scale (one week version): Change from Baseline | Baseline to week 5, 17, 23, and 29
  Tinnitus Rating Scale is a self-evaluated 11-point Likert scale assessing tinnitus loudness, annoyance, and impact on life. The scores range from 0 (no impact), to the maximum score of 10 (worst influence of the problem considered). Single scores and sum scores will be analysed.
Tinnitus Severity Scale (one week version): Change from Baseline | Baseline to week 5, 17, 23, and 29
  See outcome measure #2.
Attention and Performance Self-Assessment (ASPA) Questionnaire: Change from Baseline | Baseline to week 5, 17, 23, and 29
  The ASPA consists of 30 simple statements for which the patient can determine how regular this happens to him/her. The response options for each statement are "never", "seldom", "sometimes", "often" and "always".
Quality of Life Questionnaire (SF-36™ Health Survey): Change from Baseline | Baseline to week 17 and 29
  The SF-36 is a multipurpose health survey with 36 questions. It is a generic measure commonly used in general and specific populations, comparing the relative burden of diseases, and in differentiating the health benefits produced by a wide range of different treatments.
Hospital Anxiety and Depression Scale (HADS): Change from Baseline | Baseline to week 17 and 29
  The HADS is a self-assessment scale with 14 items which has been developed for non psychiatrists to detect states of depression and anxiety in a hospital outpatient population. Every item is rated with a scale (3= very often indeed; 2= quite often; 1= not very often; 0= not at all). Lower total scores indicate "normal", higher total scores "abnormal".

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals
Locations (75):
- United States (38):
  - Horizon Clinical Research Associates PLLC, Gilbert, Arizona
  - Phoenix Clinical, Phoenix, Arizona
  - Paradigm Clinical Research, Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - Central California Clinical Research, Fresno, California
  - UC Davis Health System, Sacramento, California
  - Colorado Otolaryngology Associates, Colorado Springs, Colorado
  - New West Physicians, Golden, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Deerpath Physicians Group, Gurnee, Illinois
  - Knight Center for Integrated Health, Peoria, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Deaconess Clinic, Inc., Newburgh, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas; Department of Otolaryngology Head & Neck Surgery, Kansas City, Kansas
  - Heartland Research Associates, LLC., Wichita, Kansas
  - Commonwealth Ear, Nose & Throat, Louisville, Kentucky
  - Glacier Ear, Nose, and Throat, Head and Neck Surgery, P.C., Kalispell, Montana
  - Immedicenter, Bloomfield, New Jersey
  - David L. Bortniker, Somerville, New Jersey
  - Erie County Medical Center, Department of Rehabilitation Medicine; State University of New York at Buffalo, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cary Medical Research, Cary, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Medical University of South Carlolina, Otolaryngology, Charleston, South Carolina
  - Austin Ear, Nose and Throat Clinic, Austin, Texas
  - Future Search Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - South Texas Research Alliance LLC, Laredo, Texas
  - Research Across America, Plano, Texas
  - Advanced Clinical Research, West Jordon, Utah
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
- Austria (4):
  - Krankenhaus der Elisabethinen, Graz
  - Bezirkskrankenhaus Kufstein, Kufstein
  - A. ö. Krankenhaus der Elisabethinen Linz, Linz
  - Clin Pharm International GmbH, Zentrum Wien, Vienna
- Brazil (7):
  - Consultório Dr. Marcelo Rates, Belo Horizonte
  - Instituto de Otorrinolaringologia Linhares, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Rio Grande
  - Faculdade de Medicina do ABC, Santo André/SP
  - Universidade Federal de São Paulo - UNIFESP, Sao Paulo/ SP
  - Instituto Ganz Sanchez, São Paulo/SP
  - Clínica OTOSUL, Valença
- Germany (12):
  - Klin. Forschung Berlin Buch GmbH, Berlin
  - Praxis im Schlosscarree, Braunschweig
  - Dr. Klaus Peter Jayme, Darmstadt
  - Dr. Christian Dörr, Dresden
  - Dr. Elisabeth Kühne, Halle
  - Dr. Werner Gieselmann, Heiligenhaus
  - Dr. Wolfgang Lotte, Iserlohn
  - ClinPharm International GmbH, Leipzig
  - HNO Praxis, Bamberger Str. 7, Lichtenfels
  - Dr. Dannesberger, Lorsch
  - LMU München, Klinikum Großhadern, München
  - Dr. Susanne Wiedemann, Nuremberg
- Mexico (14):
  - Instituto Biomédico de Investigación A.C., Aguascalientes
  - Hospital General de Chihuahua, Chihuahua City
  - Hospital Christus Muguerza del Parque, Chihuahua City
  - Clinical Research Instutute S.C., Edo. de México
  - Hospital Civil de Guadalajara "Fray Antonio Alcalde", Servicio de Otorrinolaringología; Hospital No. 278, Guadalajara Jalisco
  - Grupo Médico Terranova, Guadalajara Jalisco
  - Unidad de Investigación Clínica Cardiometábolica de Occidente S.C. (UNICAMO), Jalisco
  - Hospital General de México S.S. O.D.; Servicio de Otorrinolaringología, México D.F.
  - Hospital OCA Monterrey International Research Center (MIRC), Nuevo León
  - Hospital Universitario, Nuevo León
  - Unidad de Tratamientos Avanzados (UTRAV) S.C., Nuevo León
  - Hospital Central "Dr. Ignacio Morones Prieto"; Servicio de Otorrinolaringología, San Luis Potosí City
  - Medicentro del Parque, San Luis Potosí City
  - Unidad Médica de Especialidades del Noroeste (UMEN), Sinaloa